CLINICAL TRIAL: NCT06275022
Title: A Prospective Randomized Controlled Study on the Treatment of Cystic Lymphatic Malformation Based on Indocyanine Green-fluorescence Imaging
Brief Title: A Prospective Study on the Treatment of cLM Based on ICG Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Tao Han, Dr., Nanjing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NanjingCH011665
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Lymphatic Malformation
Keywords: indocyanine green; children; inflow; lymphography
MeSH Terms: conditions — Lymphatic Abnormalities | interventions — Sclerotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Macro/mixed cystic lymphatic A (Experimental): Inflow occlusion assisted by indocyanine green-fluorescence imaging combined with perforation of septation and sclerotherapy
  Interventions: Procedure: Inflow occlusion with perforation of septation and sclerotherapy
- Macro/mixed cystic lymphatic B (Active Comparator): Perforation of septation and sclerotherapy
  Interventions: Procedure: Perforation of septation and sclerotherapy
- Microcystic lymphatic A (Experimental): Indocyanine green-fluorescence imaging-guided partial resection and sclerotherapy
  Interventions: Procedure: Indocyanine green-guided partial resection and sclerotherapy
- Microcystic lymphatic B (Active Comparator): Partial resection and sclerotherapy
  Interventions: Procedure: Partial resection and sclerotherapy

INTERVENTIONS:
Procedure: Inflow occlusion with perforation of septation and sclerotherapy — Inflow occlusion assisted by indocyanine green-fluorescence imaging combined with perforation of septation and sclerotherapy
  Arms: Macro/mixed cystic lymphatic A
Procedure: Perforation of septation and sclerotherapy — Perforation of septation and sclerotherapy
  Arms: Macro/mixed cystic lymphatic B
Procedure: Indocyanine green-guided partial resection and sclerotherapy — Indocyanine green-fluorescence imaging-guided partial resection and sclerotherapy
  Arms: Microcystic lymphatic A
Procedure: Partial resection and sclerotherapy — Partial resection and sclerotherapy
  Arms: Microcystic lymphatic B

SUMMARY:
The goal of this prospective randomized controlled study is to explore the role of indocyanine green-fluorescence imaging in management of cystic lymphatic malformation.. To clarify the application value of indocyanine green-fluorescence imaging in both diagnosis and treatment of cystic lymphatic malformation (cLM) in children, is helpful for exploring pathogenesis of cLM, and providing a clearer scientific basis for subsequent surgical intervention. It also provides alternative for the future diagnosis and treatment of cLM.

Participants will receive indocyanine green-fluorescence imaging before operation, while the patients in control group will receive traditional operation.

Researchers will compare difference in curative effect between two groups.

ELIGIBILITY:
Inclusion Criteria:

(1) no previous intervention; (2) cLM diagnosed by pretreatment magnetic resonance imaging (MRI); (3)3 to 6 months post-treatment follow-up; (4) Superfacial cLM

Exclusion Criteria:

(1) history of iodine allergy; (2) syndromic cLM ; (3) severe liver and kidney dysfunction; (4) intralesional hemorrhage; (5) intralesional infection

Ages: 30 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 1month, 3 months
  The percentage of cured cases to total cases
Effective rate | 1 month, 3 months
  The percentage of effective cases to total cases
Treatment frequency | 3 months, 6 months
  Frequency of treatments

SECONDARY OUTCOMES:
Likert score | 6 months
  Evaluation of postoperative satisfaction
Wound infection | 1 month
  Infection of surgical region
Delayed healing | 1 month
  Delayed healing of surgical wound
Pigmentation | 1 month
  ICG-related pigmentation on skin

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Shen, Dr., Study Director — Children's Hospital of Nanjing Medical University
Locations (1):
- Children's hospital of Nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No